CLINICAL TRIAL: NCT06527118
Title: The Effect of Self-Care Education Given to Children With Educable Mental Disabilities on Children's Self-Care Skills and School Social Behaviors
Brief Title: The Effect of Self-Care Education on Self-Care Skills and School Sociality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gulendam Karsadag, Assistant Profesor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DokuzEU-HSH-GK-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Education; Intellectual Disabilities With Other Behavioral Symptoms
Keywords: Child with intellectual disabilities; self-care; socialization

STUDY DESIGN:
Intervention Model Description: pretest-posttest, follow-up control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Group to which the Self-Care Skills Learning Activity Program will be implemented (Active Comparator): The "Activity Program for Learning Self-Care Skills", which was prepared by the educator after receiving expert opinions, was applied individually to each child in the intervention group for 12 weeks. The training was 1 day a week for 40 minutes.
  Interventions: Other: ACTIVITIES TO LEARN SELF CARE SKILLS
- Self-Care Skills Learning Activity Program Not Implemented Group (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Other: ACTIVITIES TO LEARN SELF CARE SKILLS — This activity program, which was prepared to develop self-care skills, aims to teach self-care skills of children with intellectual disabilities by having fun. The program was prepared by the educator and finalized after the approval of expert opinions.
  Arms: The Group to which the Self-Care Skills Learning Activity Program will be implemented

SUMMARY:
The aim of this study is to examine the effect of self-care education given to children with educable intellectual disabilities on children's self-care skills and school social behaviors.

H1a: There is a difference between the mean scores of the children in the experimental and control groups in the "Eating Skills" subscale of the Self-Care Skills Checklist according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

H1b: There is a difference between the mean scores of the children in the experimental and control groups on the "Dressing Skills" sub-dimension of the Self-Care Skills Checklist according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

H1c: There is a difference between the mean scores of the children in the experimental and control groups on the "Personal Care Skills" sub-dimension of the Self-Care Skills Checklist according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

H1d: There is a difference between the mean scores of the children in the experimental and control groups on the "Social Competence" sub-dimension of the School Social Behavior Assessment Scale according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

DETAILED DESCRIPTION:
H1a: There is a difference between the mean scores of the children in the experimental and control groups in the "Eating Skills" subscale of the Self-Care Skills Checklist according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

H1b: There is a difference between the mean scores of the children in the experimental and control groups on the "Dressing Skills" sub-dimension of the Self-Care Skills Checklist according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

H1c: There is a difference between the mean scores of the children in the experimental and control groups on the "Personal Care Skills" sub-dimension of the Self-Care Skills Checklist according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

H1d: There is a difference between the mean scores of the children in the experimental and control groups on the "Social Competence" sub-dimension of the School Social Behavior Assessment Scale according to time (pretest, posttest, 1st follow-up, 2nd follow-up).

ELIGIBILITY:
Inclusion Criteria:

* The child has mild and moderate intellectual disability (Determined by the health reports available at the institution. Children with mild and moderate intellectual disability were included in the study).
* Between the ages of 6 and 10
* Volunteering to participate in the study and signing the informed consent form by the child's parent
* Following verbal instructions (determined by the reports given as a result of the evaluation conducted by the Guidance and Research Center)

Exclusion Criteria:

* Physical disability in addition to mental disability
* Getting sick or having an attack during work
* Illiteracy of parents

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-care Skills Checklist Scale | 12 Weeks
  "Self-Care Skills Checklist Scale" developed by Konya (2007) was used to measure children's self-care skills. The Checklist consists of 3 sections. These are Eating Skills (14 items), Dressing Skills (19 items) and Personal Care Skills (9 items). In order to determine the level of development of the skills in the checklist, "Very Adequate (5 points), Adequate (4 points), Somewhat Adequate (3 points), Inadequate (2 points), Very Inadequate (1 point)" options were used. The minimum score that can be obtained from the scale is 42 and the maximum score is 210. A high score indicates high self-care skills.
School Social Behavior Scale | 12 Weeks
  It was developed by Kenneth W. Merrell in 1993 in the United States of America as a scale that can be used by classroom teachers or other teachers in K-12 schools (from preschool to high school) to assess individual students. Cognitive-behavioral theory was used in the development of the items. The scale consists of two forms: Form A: Social Competence Form B: Negative Social Behavior Only the Social Competence Form was used in our study. In the final factor analysis of the Social Competence sub-dimension, three factors were identified: Interpersonal Relationships, Self-Control Skills and Academic Skills. The minimum score that can be obtained from the Social Competence form is 32 and the maximum score is 160. A high score indicates that the individual has high social skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No